CLINICAL TRIAL: NCT05628818
Title: Neuromodulation of Executive Dysfunction in Patients With Acute Stroke Using Transcranial Direct Current Stimulation. A Randomized-triple Blinded Controlled Clinical Trial. MODUL-EXE Trial.
Brief Title: Noninvasive Transcranial Direct Current Stimulation to Improve Executive Functions in Stroke Patients. MODUL-EXE Clinical Trial.
Acronym: MODUL-EXE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fundación Pública Andaluza para la Investigación Biomédica Andalucía Oriental (Other)
Collaborators: Instituto de Salud Carlos III (Other Government); Universidad de Almeria (Other)
Responsible Party: Principal Investigator, Laura Amaya Pascasio, Medical Doctor, investigator, Fundación Pública Andaluza para la Investigación Biomédica Andalucía Oriental
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MODUL-EXE
Record Dates: First submitted 2022-11-08; First posted 2022-11-29 (Actual); Last update posted 2023-01-18 (Actual); Status verified 2023-01

CONDITIONS: Transcranial Direct Current Stimulation
MeSH Terms: interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Anodal tDCS combined with cognitive training, stroke patients (Experimental): To stimulate the left DLPFC, the anode electrode will be placed over F3 and the cathode will be placed over the right supraorbital region (Fp2). Each stimulation will be applied for 20 min at 2mA intensity. Stimulation will be continued with the performance of three cognitive training exercises specifically designed to improving working memory, inhibitory control and cognitive flexibility.
  Interventions: Device: Transcranial Direct Current Stimulation (tDCS)
- Sham tDCS combined with cognitive training, stroke patients (Sham Comparator): To stimulate the left DLPFC, the anode electrode will be placed over F3 and the cathode will be placed over the right supraorbital region (Fp2). Each stimulation will be applied for 1 min at 2mA intensity (sham stimulation). Stimulation will be continued with the performance of three cognitive training exercises specifically designed to improving working memory, inhibitory control and cognitive flexibility.
  Interventions: Device: Sham Transcranial Direct current Stimulation

INTERVENTIONS:
Device: Transcranial Direct Current Stimulation (tDCS) — Real anodal tDCS over the left dorsolateral prefrontal cortex in acute stroke patients to improve dysexecutive syndrome. Intensity: 2 mA. Stimulation period: 20 minutes.
  Arms: Anodal tDCS combined with cognitive training, stroke patients
Device: Sham Transcranial Direct current Stimulation — Sham anodal tDCS over the left dorsolateral prefrontal cortex: anodal tDCS. Intensity: 2 mA. Stimulation period: 1 minute. Afterwards, the device will automatically shut down but the sham stimulation period will last a total of 20 minutes.
  Arms: Sham tDCS combined with cognitive training, stroke patients

SUMMARY:
This study will examine the possible effects of tDCS (Transcranial Direct Current Stimulation) treatment to the left DLPFC on executive functions in patients with an acute stroke affecting the frontal lobe or the basal ganglia. The study will include 40 acute stroke subjects. Participants will undergo a global cognitive assessment with the MoCA test and a specific assessment of executive functions with the abbreviated Wisconsin test, the five digit test and the digit span evaluation (a subtest from the Wechsler intelligence scale for adults-IV). Participants will then undergo real or sham stimulation with anodal tDCS combined with cognitive training of the main executive functions: working memory, inhibitory control and cognitive flexibility. After a 10-session intervention, a the baseline cognitive assessment will be repeated and subsequently, a follow-up of up to 12 months will be carried out.

ELIGIBILITY:
Inclusion Criteria:

* Clinical and radiological diagnosis, by means of cranial MRI or CT scan, of ischemic/hemorrhagic stroke, involving the frontal cortex or its subcortical connections (basal ganglia), in one or both hemispheres.
* The stroke occurred during the 3 months prior to inclusion in the study.
* Cognitive impairment with a dis-executive profile demonstrated by a score > 26 in the Spanish version of the MoCA test, adjusted for the number of years of formal education.
* Patients with functional independence prior to the stroke, defined as a modified rankin scale score < 3 points.
* The patient gives informed consent.

Exclusion Criteria:

* Presence of other pathologies that may be a potential cause of disability or cognitive impairment.
* Moderate or severe aphasia that hinders communication.
* Severe sensory and/or motor impairments that prevent the completion of the evaluation and/or intervention processes.
* Presence of extensive vascular leukopathia (leukoaraiosis grade 3, 4).
* History of epilepsy or seizures.
* Presence of severe systemic pathology, including cardiac, hepatic or renal failure, active neoplasia.
* Failure to meet any of the inclusion criteria recorded in the Screening for electrical stimulation of the University of Göttingen.
* Presence of:

  1. Pacemaker.
  2. Electrical and/or metallic implants.
  3. Pregnancy.
  4. Anticonvulsant medication.
  5. Tattoos in the area of electrode placement.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-02-15 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Montreal cognitive assessment | Evaluation immediately post intervention
  Global cognitive assessment test that incorporates the evaluation of executive domains such as working memory, inhibition and others such as verbal fluency, delayed recall and visuospatial capacity. Maximum score: 30. Normal if score > 26.
Montreal cognitive assessment | Evaluation post intervention: One month after intervention
  Global cognitive assessment test that incorporates the evaluation of executive domains such as working memory, inhibition and others such as verbal fluency, delayed recall and visuospatial capacity
Montreal cognitive assessment | Post intervention: Three months after intervention
  Global cognitive assessment test that incorporates the evaluation of executive domains such as working memory, inhibition and others such as verbal fluency, delayed recall and visuospatial capacity
Montreal cognitive assessment | Post intervention: Six months after intervention
  Global cognitive assessment test that incorporates the evaluation of executive domains such as working memory, inhibition and others such as verbal fluency, delayed recall and visuospatial capacity
Digit Span test | Evaluation immediately post intervention
  Evaluates working memory. Normal average reference: to have a digit span of 7 items (plus or minus 2), the greater the memory span, the better the result.
Digit Span test | Evaluation post intervention: One month after intervention
  Evaluates working memory. Normal average reference: to have a digit span of 7 items (plus or minus 2), the greater the memory span, the better the result.
Digit Span test | Post intervention: Three months after intervention
  Evaluates working memory. Normal average reference: to have a digit span of 7 items (plus or minus 2), the greater the memory span, the better the result.
Digit Span test | Post intervention: Six months after intervention
  Evaluates working memory. Normal average reference: to have a digit span of 7 items (plus or minus 2), the greater the memory span, the better the result.
Wisconsin Card Sorting Test, Brief version. | Evaluation immediately post intervention
  Assess cognitive flexibility. Respondents are required to sort numbered response cards according to different principles and to alter their approach during test administration. The global number of categories achieved will be assesed, the greater, the better the result is.
Wisconsin Card Sorting Test, Brief version. | Evaluation post intervention: One month after intervention
  Assess cognitive flexibility. Respondents are required to sort numbered response cards according to different principles and to alter their approach during test administration. The global number of categories achieved will be assesed, the greater, the better the result is.
Wisconsin Card Sorting Test, Brief version. | Post intervention: Three months after intervention
  Assess cognitive flexibility. Respondents are required to sort numbered response cards according to different principles and to alter their approach during test administration. The global number of categories achieved will be assesed, the greater, the better the result is.
Wisconsin Card Sorting Test, Brief version. | Post intervention: Six months after intervention
  Assess cognitive flexibility. Respondents are required to sort numbered response cards according to different principles and to alter their approach during test administration. The global number of categories achieved will be assesed, the greater, the better the result is.
Five digit test | Evaluation immediately post intervention
  Assessing inhibitory control. A numerical task divided into four components. The first component (reading) demands subjects to name numbers from 1 to 5 as fast as they can. On the second component (counting), they need to describe quantities from 1 to 5. The third component (choosing) involves a selective attention trial, where the subjects must not read the numbers, but rather tell how many numbers are present in each stimulus, in an incongruent condition. The last component (shifting) is similar to the choosing trial, but for each of the five stimuli, there is one previously where the subject must read the stimulus numbers. The test total scores will be used as the main measure in this study. Higher scores indicate worse performance.
Five digit test | Evaluation post intervention: One month after intervention
  Assessing inhibitory control. A numerical task divided into four components. The first component (reading) demands subjects to name numbers from 1 to 5 as fast as they can. On the second component (counting), they need to describe quantities from 1 to 5. The third component (choosing) involves a selective attention trial, where the subjects must not read the numbers, but rather tell how many numbers are present in each stimulus, in an incongruent condition. The last component (shifting) is similar to the choosing trial, but for each of the five stimuli, there is one previously where the subject must read the stimulus numbers. The test total scores will be used as the main measure in this study. Higher scores indicate worse performance.
Five digit test | Post intervention: Three months after intervention
  Assessing inhibitory control. A numerical task divided into four components. The first component (reading) demands subjects to name numbers from 1 to 5 as fast as they can. On the second component (counting), they need to describe quantities from 1 to 5. The third component (choosing) involves a selective attention trial, where the subjects must not read the numbers, but rather tell how many numbers are present in each stimulus, in an incongruent condition. The last component (shifting) is similar to the choosing trial, but for each of the five stimuli, there is one previously where the subject must read the stimulus numbers. The test total scores will be used as the main measure in this study. Higher scores indicate worse performance.
Five digit test | Post intervention: Six months after intervention
  Assessing inhibitory control. A numerical task divided into four components. The first component (reading) demands subjects to name numbers from 1 to 5 as fast as they can. On the second component (counting), they need to describe quantities from 1 to 5. The third component (choosing) involves a selective attention trial, where the subjects must not read the numbers, but rather tell how many numbers are present in each stimulus, in an incongruent condition. The last component (shifting) is similar to the choosing trial, but for each of the five stimuli, there is one previously where the subject must read the stimulus numbers. The test total scores will be used as the main measure in this study. Higher scores indicate worse performance.

SECONDARY OUTCOMES:
modified rankin scale | Evaluation immediately post intervention
  Functional assessment scale ranging from 0 (independent) to 6 (death)
modified rankin scale | Evaluation post intervention: One month after intervention
  Functional assessment scale ranging from 0 (independent) to 6 (death)
modified rankin scale | Post intervention: Three months after intervention
  Functional assessment scale ranging from 0 (independent) to 6 (death)
modified rankin scale | Post intervention: Six months after intervention
  Functional assessment scale ranging from 0 (independent) to 6 (death)
modified rankin scale | Post intervention: 12 months after intervention
  Functional assessment scale ranging from 0 (independent) to 6 (death)
Return to work | Post intervention: One month after intervention
  To determine whether the patient has been able to return to the previous job
Return to work | Post intervention: Three months after intervention
  To determine whether the patient has been able to return to the previous job
Return to work | Post intervention: 6 months after intervention
  To determine whether the patient has been able to return to the previous job
Return to work | Post intervention: 12 months after intervention
  To determine whether the patient has been able to return to the previous job
Beck's Depression Inventory | Evaluation immediately post intervention
  Evaluation of depression ranging from 0 to 63. A score > 20: significant depression (moderate-severe)
Beck's Depression Inventory | Post intervention: One month after intervention
  Evaluation of depression ranging from 0 to 63. A score > 20: significant depression
Beck's Depression Inventory | Post intervention: Three months after intervention
  Evaluation of depression ranging from 0 to 63. A score > 20: significant depression
Beck's Depression Inventory | Post intervention: Six months after intervention
  Evaluation of depression ranging from 0 to 63. A score > 20: significant depression
Apathy Evaluation Scale | Evaluation immediately post intervention
  Evaluation of presence of apathy. Consists of 18 specific items to quantify apathy within a scoring range of 18 to 72. The greater the score, the greater the apathy symptoms.
Apathy Evaluation Scale | Post intervention: One month after intervention
  Evaluation of presence of apathy. Consists of 18 specific items to quantify apathy within a scoring range of 18 to 72. The greater the score, the greater the apathy symptoms.
Apathy Evaluation Scale | Post intervention: Three months after intervention
  Evaluation of presence of apathy. Consists of 18 specific items to quantify apathy within a scoring range of 18 to 72. The greater the score, the greater the apathy symptoms.
Apathy Evaluation Scale | Post intervention: Six months after intervention
  Evaluation of presence of apathy. Consists of 18 specific items to quantify apathy within a scoring range of 18 to 72. The greater the score, the greater the apathy symptoms.
WHOQOL-BREF scale | Evaluation immediately post intervention
  Evaluation of quality of life. There are no proposed cut-off points. The higher the score, the higher the quality of life.
WHOQOL-BREF scale | Post intervention: One month after intervention
  Evaluation of quality of life. There are no proposed cut-off points. The higher the score, the higher the quality of life.
WHOQOL-BREF scale | Post intervention: Three months after intervention
  Evaluation of quality of life. There are no proposed cut-off points. The higher the score, the higher the quality of life.
WHOQOL-BREF scale | Post intervention: Six months after intervention
  Evaluation of quality of life. There are no proposed cut-off points. The higher the score, the higher the quality of life.

OTHER OUTCOMES:
Change in resting state functional connectivity | Evaluation immediately post intervention
  functional near-infrared spectroscopy-fNIRS
Change in resting state functional connectivity | Post intervention: One month after intervention
  functional near-infrared spectroscopy-fNIRS
Change in resting state functional connectivity | Post intervention: Three months after intervention
  functional near-infrared spectroscopy-fNIRS
Change in resting state functional connectivity | Post intervention: Six months after intervention
  functional near-infrared spectroscopy-fNIRS
Motor evaluation | Evaluation immediately post intervention
  Nine-hole peg test and Timed 25-Foot Walk tests as motor status monitoring tasks
Motor evaluation | Post intervention: One month after intervention
  Nine-hole peg test and Timed 25-Foot Walk tests as motor status monitoring tasks
Motor evaluation | Post intervention: Three months after intervention
  Nine-hole peg test and Timed 25-Foot Walk tests as motor status monitoring tasks
Motor evaluation | Post intervention: Six months after intervention
  Nine-hole peg test and Timed 25-Foot Walk tests as motor status monitoring tasks
Blood biomarkers | Evaluation immediately post intervention
  Brain-derived neurotrophic factor (BDNF), glial cell-derived neurotrophic factor (GDNF), nerve growth factor (NGF), pituitary adenylate cyclase polypeptide 38 (PACAP-38), insulin-like growth factor type 1 (IGF-1), interleukins 2, 4, 6, 8 and 10; and tumour necrosis factor (TNF).

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Martinez Sanchez, PhD, Principal Investigator — Torrecardenas University Hospital; Pilar Flores Cubos, Professor, PhD, Study Director — Department of Psychology. University of Almeria
Locations (1):
- Torrecardenas University Hospital, Almería, Almeria, Spain

IPD SHARING:
Plan to Share IPD: Yes